CLINICAL TRIAL: NCT01334190
Title: A Prospective Observational Study of the Performance of Zarin in Kenya
Status: Completed | Type: Observational
Sponsor: FHI 360 (Other)
Collaborators: United States Agency for International Development (USAID) (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: 10264
Record Dates: First submitted 2011-04-11; First posted 2011-04-13 (Estimated); Last update posted 2013-07-02 (Estimated); Status verified 2013-07

CONDITIONS: Contraceptive Usage
Keywords: AE adverse event; AIDS acquired immunodeficiency syndrome; ALT (SGPT) alanine aminotransferase; ART antiretroviral therapy; AST (SGOT) aspartate aminotransferase; DCF data collection forms; DMC Data Monitoring Committee; FDA (U.S.) Food and Drug Administration; GCP Good Clinical Practice guidelines; HB sAg Hepatitis B surface antigen; ICH International Conference of Harmonisation; IND Investigational New Drug Application; IRB Institutional Review Board; IU international units; mg milligram(s); mm3 cubic millimeter(s); PCR polymerase chain reaction; SAE serious adverse event; µg microgram; ULN upper limit of the normal range; WB Western Blot; post-marketing monitoring; safety; efficacy; acceptability
MeSH Terms: conditions — Contraception Behavior; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

SUMMARY:
This will be a non-comparative prospective observational study of women using Zarin as a primary method of contraception in Kenya. It will be conducted in close collaboration with the Kenya MoH in several MoH-affiliated clinics that have experience with implants and sufficient expected flow of implant users per month. The investigators will enroll a total of 600 women divided into two cohorts in this one-year prospective study:

* a prospective cohort consisting of 300 women who will be followed-up 3 and 12 months after enrollment; and
* a surveillance cohort of 300 women who will report back to the clinic during 12 months after enrollment only if they have complications, medical problems, pregnancy, or want to remove the implant

The main study outcomes are pregnancy, immediate and delayed complications associated with insertion or removal, adverse events, early discontinuation and reasons for discontinuation, and level of women's satisfaction with Zarin services.

DETAILED DESCRIPTION:
A non-comparative prospective observational study of women using Zarin as a primary method of contraception in Kenya. It will be conducted in close collaboration with the Kenya MoH in several MoH-affiliated clinics that have experience with implants and sufficient expected flow of implant users per month. The investigators will enroll a total of 600 women divided into two cohorts in this one-year prospective study:

* a prospective cohort consisting of 300 women who will be followed-up 3 and 12 months after enrollment; and
* a surveillance cohort of 300 women who will report back to the clinic during 12 months after enrollment only if they have complications, medical problems, pregnancy, or want to remove the implant

The main study outcomes are pregnancy, immediate and delayed complications associated with insertion or removal, adverse events, early discontinuation and reasons for discontinuation, and level of women's satisfaction with Zarin services.

ELIGIBILITY:
Inclusion Criteria:

* be aged 18-44 years, inclusive
* be willing to sign an informed consent document
* be willing to give contact information for follow up
* agree to return for follow-up visits
* have decided to receive Zarin as a method of contraception and met the clinic criteria for eligibility of this method of contraception

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: healthy women aged 18-44
Sampling Method: Non-Probability Sample
Enrollment: 602 (Actual)
Dates: Start 2011-06; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
The cumulative probability of pregnancy | 1 year

SECONDARY OUTCOMES:
Prevalence and incidence rates of immediate and delayed complications associated with insertion or removal | 1 year
Prevalence and incidence rate of adverse events | 1 year
The cumulative probability of early discontinuation of Zarin through one year | 1 year
Reasons for discontinuation | 1 year
Level of women's satisfaction with Zarin services | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Vera Halpern, MD, Principal Investigator — FHI 360
Locations (1):
- FHI, Nairobi, Nairobi County, Kenya